CLINICAL TRIAL: NCT04170166
Title: Subacromial Injections for Shoulder Subacromial Pain Syndrome - Comparing Anterolateral Versus Posterior Approach: A Randomised Controlled Trial
Brief Title: Subacromial Injections for Shoulder Subacromial Pain Syndrome - Anterolateral vs Posterior Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blackpool Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Charalambos Charalambous, Consultant Orthopaedic Surgeon, Blackpool Teaching Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 249246
Record Dates: First submitted 2019-10-30; First posted 2019-11-20 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Shoulder Subacromial Pain Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterolateral Approach (Active Comparator): The randomised group of patients receiving the subacromial steroid injection via an anterolateral approach
  Interventions: Procedure: Anterolateral subacromial steroid injection
- Posterior Approach (Active Comparator): The randomised group of patients receiving the subacromial steroid injection via a posterior approach
  Interventions: Procedure: Posterior subacromial steroid injection

INTERVENTIONS:
Procedure: Anterolateral subacromial steroid injection — Applying to the anterolateral approach arm, this group will receive their subacromial steroid injection via an anterolateral approach
  Arms: Anterolateral Approach
Procedure: Posterior subacromial steroid injection — Applying to the posterior approach arm, this group will receive their subacromial steroid injection via an posterior approach
  Arms: Posterior Approach

SUMMARY:
This study aims to determine if there is any difference in terms of pain relief in patients with shoulder subacromial pain syndrome, when given a steroid injection into the subacromial space via an anterolateral approach compared to a posterior approach.

DETAILED DESCRIPTION:
Patients who present with subacromial pain syndrome (disorders such as subacromial bursitis, rotator cuff tendinopathy, calcific tendinitis, subacromial inflammation with a partial thickness rotator cuff tear) to the orthopaedic outpatient clinic are treated initially with a subacromial steroid injection in addition to physiotherapy for a period of 3 months. This applies to patients who have had no other treatments previously as well as to patients who have had previous physiotherapy or steroid injections prior to presentation. Patients who do not want to undergo the treatment offered are either treated with simple analgesia, sole physiotherapy or surgery.

When a patient with one of the above conditions agrees to go ahead with a steroid injection followed by physiotherapy, the steroid injection is given at the earliest opportunity. The steroid injection is given into the subacromial space either using the anterolateral (front-side) approach (1 cm below and behind the anterior edge of the acromion with the needle aiming towards the under surface of the acromion) or using the posterior (back-side) approach ( 1cm inferior and medial to the posterlateral acromial edge with the needle pointing towards the anterolateral aspect of the acromion). The exact approach is determined according to the preference of the person carrying out the injection. As a routine we use a 10ml syringe containing 10mls of 0.25% Marcaine along with 40mg triamcinolone with an 18 gauge (green) needle. It is normal for patients to complain of some discomfort during the injection. If a patient experiences any significant discomfort or they cannot tolerate the injection for whatever reason, then the injection is discontinued and is not reattempted using a different approach.

Following the injection, patients are questioned on any discomfort experienced during the injection and on whether or not their pain has improved. They are then taken through a protocol of physiotherapy for their shoulder over the subsequent 3 months. A protocol is issued for guidance however therapists are allowed to use other modalities as per their discretion. The frequency of appointments with physiotherapy will depend on patient's symptoms as well as their progression. For study purposes a frequency record of these meetings will be kept and matched to the overall OSS. Patients are seen routinely in 3 months following an injection in order to assess any improvement in symptomatology using the OSS, visual analogue score, DASH and SF36 questionaires. If the symptoms have improved then no further intervention is taken. Further OSS, visual analogue pain score, DASH and SF36 questionaires will be posted out at 6 months and 1 year. On the other hand, if they are still troubled with symptoms then the possibility of further injections or surgery is discussed.

The aim of this study is to compare the two approaches that are currently used for subacromial steroid injections, namely the anterolateral and posterior approach, with regards to their effectiveness in improving shoulder symptoms. There will be no deviation from our routine protocol other than randomising patients who agree to participate in this study to either the anterolateral or posterior approach.

In summary, it is patients who are seen in clinic with a subacromial pathology and subsequently diagnosed with shoulder subacromial pain syndrome, who are offered an injection. Those who agree to have an injection will then be invited to participate in the study. An information leaflet will be given to all potential participants and they will be allowed sufficient time to read through it, digest all the information and ask any questions they may have before making a decision regarding their participation. Those who agree to participate will be randomly allocated, using sealed envelopes to one of the two approaches for the injection. The injection will then be administered via the selected approach by a clinician who is qualified in carrying out the procedure. Patients will be asked about any discomfort experienced during the injection, improvement in pain following the injection prior to leaving hospital and overall satisfaction with the injection. Following this patients will have physiotherapy as an outpatient as routine and will be seen at about 3 months post injection for a further assessment at the clinic. Again the shoulder assessment will be repeated on that occasion. Shoulder assessment questionaires will be posted out for completion at 6 months and 1 year (OSS, pain on visial analogue scale, DASH and SF36) There will be no change in patients care from routine practice other than the randomisation of the approach used for the injection. Patients who are invited to participate in the study and agree to participate will have their GP informed of their participation.

Assessments

1. Prior to injection: assessment of pain using a visual analogue score, clinical assessment of shoulder movement and completion of a modified Oxford Shoulder Score, Disabilities of Shoulder, Arm and Hand questionaires and Short Form 36 Health Survey.
2. 20-30 minutes Post injection: assessment of pain using a visual analogue score
3. Prior to leaving hospital: pain experienced during the administration of the injection and the overall satisfaction with the injection
4. 3 months post injection: assessment of pain using a visual analogue score, clinical assessment of shoulder movement and completion of a modified Oxford Shoulder Score, Disabilities of Shoulder, Arm and Hand questionaires and Short Form 36 Health Survey.
5. 6 months and 1 year post injection: assessment of pain using visual analogue score and completion of a modified Oxford Shoulder Score, Disabilities of Shoulder, Arm and Hand questionaires and Short Form 36 Health Survey via post.

The main outcome for this study will be the Oxford Shoulder Score (OSS) at 3 months post-injection. In addition to the standard OSS, the questionnaire will inquire about general symptoms and signs, duration, hand dominance, previous injuries to the shoulder and previous treatments to the shoulder. The follow up questionnaire will be identical to the initial questionnaire but excluding questions on previous treatments, hand dominance, injuries and duration.

Other demographics that will be recorded on the pre-designed pro forma include: number and frequency of physiotherapy sessions pre and post injection, and subsequent need for further management.

Hard copies of data (questionnaires and forms) collected will be placed into the patient's notes. At the same time this data will be recorded electronically on an Excel database and saved on an encrypted, password protected memory stick. This memory stick will be stored in a locked filing cabinet in the orthopaedic department at Blackpool Victoria Hospital. Please note: The electronic data will contain NO identifiable information. Participants will be identified by a unique study I.D number which can only be linked to them by members of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with shoulder subacromial pain syndrome
* Age ≥ 18
* Capacity to give valid consent for participation
* Able to complete the follow up

Exclusion Criteria:

* Age < 18
* Lacking capacity/unable to give valid consent for participation
* Full thickness rotator cuff tear diagnosed on either Ultrasound scan or Magnestic Resonance Imaging
* Unable to complete follow up
* Unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 3 months
  The primary outcome measure will be the change in the Oxford Shoulder Score at 3 months post injection. Scores range from 0-48 with 48 being the best possible outcome.

SECONDARY OUTCOMES:
Oxford Shoulder Score | 6 months and 1 year
  Change in the Oxford Shoulder Score at 6 months and 1 year post injection. Scores range from 0-48 with 48 being the best possible outcome.
Pain on visual analogue scale | 3 months, 6 months and 1 year post injection
  Change in pain on the visual analogue scale at 3 months, 6 months and 1 year post injection. As this is a visual analogue scale this is a visual scale with no numeric values attached however on the left side of the scale will be no pain and the right side will be maximal pain.
Disabilities of Arm, Shoulder and Hand Questionnaire | 3 months, 6 months and 1 year
  Change in the Disabilities of Arm, Shoulder and Hand Questionnaire score at 3 months, 6 months and 1 year post injection. This is a score that ranges from 0-100 with 0 meaning no disability and 100 meaning most severe disability.
Short Form 36 Health Survey Score | 3 months, 6 months and 1 year
  Change in the Short From 36 Health Survey Score at 3 months, 6 months and 1 year post injection. This is a range from 0-100 with the higher the score, the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Charalambous, Principal Investigator — Consultant Orthopaedic Surgeon
Locations (1):
- Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, United Kingdom

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04170166/Prot_SAP_ICF_000.pdf